CLINICAL TRIAL: NCT06765733
Title: The Study of Safety and Preliminary Efficacy of Aleeto in Patients With MultIple System Atrophy
Acronym: SPRITE
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, yilong Wang, Vice President of Beijing Tiantan Hospital, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2024-314-02
Record Dates: First submitted 2024-11-26; First posted 2025-01-09 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Multiple System Atrophy - Parkinsonian Subtype (MSA-P); Multiple System Atrophy, MSA
Keywords: Multiple System Atrophy; Treatment; Exosomes; Neurorepair
MeSH Terms: conditions — Multiple System Atrophy; Thyroid Dyshormonogenesis 2A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Intrathecal administration combined with intravenous administration of Aleeto of Aleeto was given to each MSA patient in the intervention group, with intrathecal administration on days 1, 31 and 61 and intravenous administration on days 2 to 14, 32 to 44±3 and 62 to 74±5, and treatment was given once a day.
  intrathecal administration: 8 mL sodium chloride injection + Aleeto (130 μg/branch) for intrathecal administration, which was completed in about 5 minutes; intravenous administration: Aleeto (130 μg/branch) was dissolved in 100 ml sodium chloride injection, which was completed in about 30-40 minutes. After completion of the above treatments and 90±7 days of follow-up, all subjects entered the OLE study phase. During this period, all participants were given the option of continuing to receive 3 phases (on Days 91 to 104±7, Days 121 to 134±7, and Days 151 to 164±7) of intravenous Aleeto administration (14 consecutive days of Aleeto 130 μg qd i.v. in each phase).
  Interventions: Drug: Aleeto
- Control group (No Intervention): Each MSA patient in the blank control group received only basic treatment with no trial-related treatment.
  After completion of the above treatments and 90±7 days of follow-up, all subjects entered the OLE study phase. During this period, all participants were given the option of continuing to receive 3 phases (on Days 91 to 104±7, Days 121 to 134±7, and Days 151 to 164±7) of intravenous Aleeto administration (14 consecutive days of Aleeto 130 μg qd i.v. in each phase).

INTERVENTIONS:
Drug: Aleeto — "Aleeto" is a nerve repair protein developed by Darwin Start (Beijing) Biopharmaceutical Co., Ltd. It is a group of specific microenvironmental protein polymers secreted under the emergency conditions of stem cells. It has the advantages of selective assembly, targeted delivery, efficient repair of damaged tissues, high safety, chemical stability, easy storage, etc., and has a powerful neural repair function. According to the groups, patients would be treated with Aleeto via intrathecal injection or intravenous injection.
  Arms: Intervention group

SUMMARY:
This is a single-center, prospective, randomized, open-label, blinded outcome assessment (PROBE) study. At the end of the PROBE study, patients who have completed the study may opt to enter the open-label extension (OLE) study. The objective of the study is to evaluate the safety, tolerability and potential preliminary efficacy of Aleeto in the treatment of patients with multiple system atrophy (MSA).

DETAILED DESCRIPTION:
Multiple system atrophy (MSA) is a progressive neurodegenerative disorder characterized by a blend of autonomic dysfunction, Parkinson's syndrome, and cerebellar syndrome. The incidence of MSA ranges from 1.9 to 4.9 per 100,000 individuals, with an average age of onset of 56.2 years. Among individuals aged 50 years and older, the prevalence stands at 3.0 per 100,000. The mean age of MSA onset is 56.2 years, and the median survival ranges from 6.2 to 7.5 years. Severe autonomic dysfunction manifests early in the disease course, impacting patient survival. The challenges in early diagnosis, rapid disease progression, and bleak prognosis of MSA lead to approximately half of patients needing a walker or assistance from family members for mobility within three years of motor symptom onset. By the fifth year, 60% of patients rely on a wheelchair, and the majority become bedridden within six to eight years. This progression significantly diminishes their quality of life and survival.

Treating MSA, a rare neurodegenerative condition, remains a significant challenge. Current symptomatic and supportive therapies fall short of meeting the treatment requirements of MSA patients. Furthermore, potential adverse effects and disease progression factors restrict the use of certain drugs, highlighting the critical need for the development of disease-modifying or neuroprotective agents to decelerate disease advancement.

"Aleeto, a nerve repair protein created by Darwin Origin (Beijing) Biopharmaceutical Co.LTD, is derived from cellular exosomes, a set of specific microenvironmental protein polymers secreted by stem cells under emergency conditions. It boasts selective assembly, targeted delivery, highly efficient tissue repair, exceptional safety, chemical stability, and convenient storage. Previous basic research has indicated Aleeto's potential for promoting endogenous neural tissue repair, exhibiting significant neuroprotective and neurorestorative effects in animal models. Consequently, this project initiates a single-center, prospective, randomized, open-label, blinded outcome assessment (PROBE) study, followed by an open-label extension (OLE) study. The objectives are to evaluate the safety, tolerability, and potential preliminary efficacy of Aleeto in treating MSA patients and to explore effective MSA treatments.

This study aims to recruit 20 MSA-parkinsonian type (MSA-P) patients aged between 30 and 75 years. The visit content at each stage of this study includes vital signs, neurological examination, laboratory tests (such as routine blood test, blood biochemical examination, coagulation test, etc.), imaging examinations (such as MRI, bladder ultrasound), neurological assessments (such as unified multiple system atrophy rating scale [UMSARS], composite autonomic symptom score [COMPASS], EuroQol Five Dimensions Questionnaire [EQ-5D], Mini-Mental State Examination [MMSE]), and cerebrospinal fluid collection. Different stages of the study focus on monitoring patients' concomitant medications, adverse events, and serious adverse events. Detailed follow-up is conducted at the end of each treatment period, with face-to-face visits at specific time points. Additionally, researchers are required to promptly report and manage events when patients develop new neurological symptoms or suspicious events. The follow-up content of the study includes treatment and follow-up assessments at multiple stages. Initially, comprehensive physical examinations, laboratory tests (including blood, urine, pregnancy tests, etc.), multidimensional scoring assessments (such as UMSARS, COMPASS, EQ-5D, MMSE), and brain examinations through imaging techniques such as 3T MRI are performed on subjects at baseline. Subsequently, subjects enter three treatment periods and follow-up stages lasting a total of 90 days, with daily monitoring of vital signs, cerebrospinal fluid collection, laboratory tests, and adverse event documentation in each stage. Follow-up during the Open-Label Extension (OLE) phase (from day 90 to day 165 post-randomization) continues monitoring of vital signs, laboratory tests, and adverse event recording. At the follow-up visits on day 90, day 180, and day 360, comprehensive physical examinations, laboratory tests, gait analysis, bladder ultrasound, MRI, and repeat UMSARS, COMPASS, EQ-5D scoring are conducted. Additionally, if patients experience new neurological symptoms or suspicious events, additional visits will be carried out, and researchers are required to submit and interpret relevant data within 72 hours of the event occurrence.

The protocol of this study has been approved by the Ethics Committee of Beijing Tiantan Hospital. All participants will provide written informed consents before entering the study.

ELIGIBILITY:
Inclusion Criteria:

1.30 years ≤ 75 years of age, regardless of sex; 2.Clinically confirmed or clinically probable MSA-P; 3.Poor response to levodopa; 4.MSA-related motor symptom onset ≤5 years at first visit; 5.Walking ≥10 meters independently or with a walking aid; 6.Expected survival of ≥1 year, as determined by the investigator; 7.Signed informed consent.

Exclusion Criteria:

1. Head MRI at screening showing evidence of other CNS lesions consistent with a diagnosis of neurodegenerative disease other than MSA;
2. Patients with MMSE scores indicative of dementia prior to enrolment (≤17 points for illiterate individuals, ≤20 points for individuals with elementary school education, ≤24 points for individuals with junior high school education or higher) or those with a prior confirmed diagnosis of dementia;
3. Head MRI at screening showing other significant pathological findings including but not limited to: cerebral hemorrhage, acute phase of cerebral infarction, aneurysm, vascular malformation, infectious lesion, brain tumor or other space-occupying lesion (meningiomas or arachnoid cysts with a maximum diameter of <1 cm need not be excluded);
4. Presence of immune disorders that are inadequately controlled or require treatment with biological agents;
5. Known history of allergy to biological agents such as proteins and cell products;
6. Patients who have received any vaccination within 1 month;
7. Patients with pre-existing, clearly diagnosed malignant tumor or being treated with anti-tumor drugs;
8. Patients with a history of clearly diagnosed epilepsy or taking antiepileptic drugs;
9. Presence of lumbar spine disease and deformity or other contraindications to lumbar puncture;
10. Patients with abnormal coagulation function prior to enrolment (e.g., platelet count <100 × 10E9/L; prothrombin time [PT] >3 s), previous diagnosis of coagulation disorders such as hemophilia, and patients currently receiving more than two types of antiplatelet medication;
11. Contraindications to MRI (e.g. claustrophobia, internal placement of pacemakers or paramagnetic metals, etc.);
12. With severe hepatic insufficiency, renal insufficiency or severe cardiac insufficiency (severe hepatic insufficiency refers to ALT value≥2.0 times the upper limit of normal value or AST value≥2.0 times the upper limit of normal value; severe renal insufficiency refers to CRE≥1.5 times the upper limit of normal value or eGFR<40mL/min/1.73m2; severe cardiac insufficiency refers to NYHA class 3-4);
13. Hepatitis B active infection (hepatitis B surface antigen positive and/or serum HBV DNA positive or serum HBV DNA > 2 × 10E8 IU/ml;
14. Hepatitis C virus antibody positive or history of positive test;
15. Positive HIV test or history of positive test;
16. Patients with a combined history of alcohol or drug abuse or alcohol or drug dependence within 2 years;
17. Other psychiatric disorders diagnosed according to DSM-V diagnostic criteria, or significant suicide intent;
18. Patients who are pregnant, breast-feeding, or who are likely to become pregnant and plan to become pregnant;
19. Patients who are participating in other interventional studies or using other investigational biological agents, drugs, or devices, and patients who have used other experimental drugs within 1 month or within 5 drug half-lives;
20. Unable to be cooperative and complete the follow-up due to other reasons.
21. Patients who, in the opinion of the investigator, are not suitable for participation in this trial.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-31 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of investigator-reported adverse events (AEs) and serious adverse events (SAEs) | Day 90±7 after randomization
  Incidence of investigator-reported adverse events (AEs) and serious adverse events (SAEs) within 90±7 days after randomization;
The incidence of changes in clinical laboratory test parameters, changes in vital signs, neurological examination abnormalities and ECG abnormalities | Day 90±7 after randomization
  Laboratory tests include: routine blood test, coagulation test, blood biochemical examination, urinalysis (note that abnormal changes in laboratory test results may need to be reviewed to further determine and assess their relevance to the study). Vital signs include: abnormal body temperature (≥38℃ or ≤35℃), blood pressure (systolic blood pressure ≥180mmHg or <90mmHg), respiration (>24 beats/min and other rhythm abnormalities), heart rate (>100%), and blood pressure (<10%).

SECONDARY OUTCOMES:
Changes in the unified multiple system atrophy rating scale (UMSARS) part scores, sum of part 1 and 2 scores | Day 15, 45±3, 75±5 and 90±7 after randomization
  The unified multiple system atrophy rating scale (UMSARS) is composed of four subscales: UMSARS-I (12 items) rates patient-reported functional disability, UMSARS-II (14 items) assesses motor impairment based on a clinical examination, UMSARS-III records blood pressure and heart rate in the supine and standing positions, and UMSARS-IV (1 item) rates chore-based disability. Higher scores on the UMSARS indicate greater disability.
Changes in the composite autonomic symptom score (COMPASS) scores | Day 15, 45±3, 75±5 and 90±7 after randomization
  The Composite Autonomic Symptom Score (COMPASS) is a revised version of the 169-item Autonomic Symptom Profile assessing 11 domains of autonomic function, to the 31-item COMPASS, now assessing six domains: orthostatic hypotension (maximum score 10), vasomotor (maximum score 6), secretomotor (maximum score 7), gastrointestinal (maximum score 28), bladder (maximum score 9), and pupillomotor functions (maximum score 15). Scores from each component are recorded and a weighted total score is calculated. Higher scores on this scale indicate more severe clinical symptoms related to autonomic dysfunction. It is a validated, easy-to-use self-assessment instrument designed for clinical autonomic research and practice.
Changes in the incidence of orthostatic hypotension | Day 15, 45±3, 75±5 and 90±7 after randomization
  Changes in the incidence of orthostatic hypotension in patients on days 8, 38±3, 68±5, and 90±7 after randomization as measured by recumbent-upright blood pressure monitoring/24-hour ambulatory blood pressure monitoring/head-upright tilt test;
Variation of three-dimensional gait analysis parameters under multitasking | Day 90±7 after randomization
  Changes in three-dimensional gait analysis parameters under multitasking in patients on day 90±7 after randomization;
EuroQol Five Dimensions Questionnaire (EQ-5D) | Day 90±7 after randomization
  The EuroQol Five Dimensions Questionnaire (EQ-5D) consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Changes in the Berg Balance Scale | Day 90±7 after randomization
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete.
Changes in the Fatigue Severity Scale (FSS) | Day 90±7 days after randomization
  The Fatigue Severity Scale (FSS) evaluates impact of fatigue through a short self-report questionnaire consisting in statements that help the patient rate the severity of their fatigue symptoms as related to fatigue impact on their daily activities and lifestyle. The sum of the 9 items is then divided by 9 to obtain the average response value, hence the FSS ranges from 1 to 7. The higher the score, the greater the severity of fatigue and the negative effect on the person's activities.
Changes in the Zung Self - Rating Anxiety Scale (SAS) | Day 90±7 days after randomization
  The Zung Self-Rating Anxiety Scale (SAS) is a psychological assessment tool designed to quantify a person's level of anxiety. It consists of 20 items, each of which is scored on a four-point scale ranging from "none or a little of the time" to "most or all of the time." This self-administered questionnaire is utilized in both clinical and research settings to evaluate the presence and intensity of anxiety symptoms.
Changes in the Zung Self-Rating Depression Scale | Day 90±7 days after randomization
  The Zung Self-Rating Depression Scale was designed by W.W. Zung to assess the level of depression for patients diagnosed with depressive disorder. The Zung Self-Rating Depression Scale is a short self-administered survey to quantify the depressed status of a patient. There are 20 items on the scale that rate the four common characteristics of depression: the pervasive effect, the physiological equivalents, other disturbances, and psychomotor activities. There are ten positively worded and ten negatively worded questions. Each question is scored on a scale of 1-4 (a little of the time, some of the time, good part of the time, most of the time).
Changes in immunological indices (lymphocyte subpopulation) | Day 15, 30±3, 45±3, 60±5, 75±5, 105±7, 135±7, and 165±7 after randomization
  Changes in immunological indices (lymphocyte subpopulation) on days 15, 30±3, 45±3, 60±5, 75±5, 105±7, 135±7, and 165±7 after randomization.

OTHER OUTCOMES:
Changes in postvoid residual urine volume (bladder ultrasound) in patients; | Day 90±7 after randomization
  Changes in postvoid residual urine volume (bladder ultrasound) in patients on day 90±7 after randomization;
Changes in plasma biomarkers (NFL, α-syn, Tau protein, Aβ40/42/43, YKL-40, CoQ10, UA, Hcy, and other biomarkers) associated with neural repair, vascular endothelial injury, inflammatory factors and histology | Day 15, 30±3, 60±5, 90±7, 180±14, and 360±14 after randomization
  Changes in NFL, α-syn, Tau protein, Aβ40/42/43, YKL-40, CoQ10, UA, Hcy, and other biomarkers related to neural repair, vascular endothelial injury, inflammatory factors, and histology in plasma on days 15, 30±3, 60±5, 90±7, 180±14, and 360±14 after randomization;
Changes in plasma biomarkers (NFL, α-syn, Tau protein, Aβ40/42/43, YKL-40, CoQ10, UA, Hcy, and other biomarkers) associated with neural repair, vascular endothelial injury, inflammatory factors and histology | Day 31±3 and 61±5 after randomization
  Changes in NFL, α-syn, Tau protein, Aβ40/42/43, YKL-40, CoQ10, UA, Hcy, and other biomarkers related to neural repair, vascular endothelial injury, inflammatory factors, and histology in plasma on days 31±3 and 61±5 after randomization;
Changes in patients' 3T MRI imaging features (degree of cerebral atrophy in the putamen, other brain regions and whole brain; iron deposition; image parameters of diffusion tensor imaging; etc.) | Day 90±7 after randomization
  3T MRI imaging features: degree of cerebral atrophy in the putamen, other brain regions and whole brain; iron deposition assessed by quantifying magnetic susceptibility values through the use of quantitative susceptibility mapping; image parameters of diffusion tensor imaging, including mean diffusivity and fractional anisotropy.
Changes in patient's blood oxygen-level-dependent functional magnetic resonance imaging (BOLD fMRI) | Day 90±7 after randomization
  Changes in patient's blood oxygen-level-dependent functional magnetic resonance imaging (BOLD fMRI) at day 90±7 after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wang, M.D., Principal Investigator — Beijing Tiantan Hospital, Capital Medical University, Beijing, China; Tao Feng, M.D., Principal Investigator — Beijing Tiantan Hospital, Capital Medical University, Beijing, China
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No